CLINICAL TRIAL: NCT00866216
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Geneva 600mg Azithromycin Monohydrate Tablets and Pfizer Inc. (Zithromax) 600mg Azithromycin Dihydrate Tablets in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: Comparative Bioavailability Study of 600mg Azithromycin Monohydrate Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D., VP Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA02511
Record Dates: First submitted 2009-03-18; First posted 2009-03-20 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Azithromycin

ARMS (2):
- 1 (Experimental): Azithromycin Monohydrate 600mg Tablets
  Interventions: Drug: Azithromycin Monohydrate 600mg Tablets Geneva Pharmaceuticals
- 2 (Active Comparator): Zithromax (Azithromycin Dihydrate) 600mg Tablets
  Interventions: Drug: Zithromax (Azithromycin Dihydrate) 600mg Tablets Pfizer Inc.

INTERVENTIONS:
Drug: Azithromycin Monohydrate 600mg Tablets Geneva Pharmaceuticals
  Arms: 1
Drug: Zithromax (Azithromycin Dihydrate) 600mg Tablets Pfizer Inc.
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence of Azithromycin Monohydrate 600 mg Tablets.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on physical exam, medical history, or clinical laboratory results on screening

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C
* Treatment for drug or alcohol dependence
* Female subjects who are pregnant or lactating

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2003-08; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 32 days

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Marion, Principal Investigator — MDS Pharma